CLINICAL TRIAL: NCT07328789
Title: Assessment of the Effectiveness of Comprehensive Cardiac Rehabilitation and Identification of Factors Modulating Its Results
Brief Title: Factors Influencing Cardiac Rehabilitation Success
Status: Not yet recruiting | Type: Observational
Sponsor: Pomeranian Medical University Szczecin (Other)
Responsible Party: Principal Investigator, Aleksandra Rył, Clinical Professor, Pomeranian Medical University Szczecin
Other Study IDs: KB-006/65/2025
Record Dates: First submitted 2025-12-01; First posted 2026-01-09 (Actual); Last update posted 2026-01-09 (Actual); Status verified 2025-12

CONDITIONS: Rehabilitation
Keywords: Cardiac Rehabilitation; Sex Hormones; Cognitive Dysfunction
MeSH Terms: conditions — Cognitive Dysfunction

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Rehabilitation effective — This study is an observational, non-pharmacological, multi-domain assessment of patients undergoing standard comprehensive cardiac rehabilitation (CR) following CABG surgery. The intervention involves a detailed, longitudinal, three-stage evaluation (Baseline, Post-Rehab, 3-6 Month Follow-up) of the factors influencing CR outcomes.
  The CR itself is a standard hospital-based program, but the research intervention is distinguished by its holistic focus on measuring and correlating:
  Objective Functional Data: Exercise capacity (6MWT), muscle strength, diaphragm function (USG), and postural stability.
  Multifactorial Co-morbidities: Screening for Obstructive Sleep Apnea (OSA) (NOX-T3), Cognitive Dysfunction (MoCA/MMSE), and the role of oral health in OSA risk.
  Biological & Hormonal Profile: Measuring Sex Hormones (Testosterone, Estradiol) and Myokines (Irisin, Myostatin) to understand personalized metabolic and adaptive responses to the rehabilitation program.
  The intervention aims to

SUMMARY:
Cardiovascular diseases, especially after life-saving surgeries, require comprehensive cardiac rehabilitation (CR). We know that the effectiveness of CR varies among patients. The main goal of this study is to understand which factors-psychological, physical, cognitive, biochemical, and hormonal-influence the success and long-term durability of the recovery process. These findings will help us create more effective and personalized treatment programs.

Who is Being Studied and What is Being Assessed? Study Group: 150 patients of both sexes, aged 50-80 years, hospitalized in the cardiac rehabilitation ward, primarily after Coronary Artery Bypass Grafting (CABG).

Study Period: Patients will be assessed at the start of their hospital stay, at the end of rehabilitation, and again 3-6 months after discharge.

Key Assessment Areas (Modulating Factors)

Physical Status and Fitness:

Exercise tolerance (6-Minute Walk Test).

Muscle strength (handgrip), balance, and gait.

Body composition (analysis of muscle mass and fat tissue).

Respiratory function and diaphragm mobility (ultrasound).

Psychological and Cognitive Factors:

Assessment of anxiety, depression, and general mental well-being.

Evaluation of cognitive functions (memory, concentration) following cardiac surgery.

Sleep Problems (OSA):

Assessment of the risk and severity of Obstructive Sleep Apnea (OSA), which is common in cardiac patients.

Analysis of OSA risk factors related to oral health (dentition, microbiome) and craniofacial structure.

Biological Markers:

Hormonal tests (e.g., testosterone, estradiol) and their correlation with psycho-physical condition and the rehabilitation process.

Analysis of metabolic and muscle-related biomarkers (e.g., myokines: irisin, myostatin).

DETAILED DESCRIPTION:
Cardiovascular diseases, particularly advanced coronary artery disease requiring interventions like Coronary Artery Bypass Grafting (CABG), are major global health concerns. Comprehensive cardiac rehabilitation (CR) is a crucial element in patient recovery, yet its effectiveness varies significantly. The main objective of this project is the comprehensive evaluation of the actual effectiveness of standard CR and the identification of multi-faceted factors-biological, functional, and psychosocial-that influence its outcomes and long-term prognosis.

Methodology and Study Design The project plans to recruit 150 male and female patients, aged 50-80 years, who are hospitalized in the cardiac rehabilitation ward, primarily following CABG surgery.

Assessments will be conducted at three key time points to monitor the dynamic nature of changes:

Baseline (T0): At the beginning of cardiac rehabilitation.

Post-Rehab (T1): At the conclusion of the standard rehabilitation program.

Follow-up (T2): Approximately 3-6 months after the patient's discharge.

Detailed Research Domains

The study will focus on several key domains to comprehensively assess the mechanisms underlying recovery:

A. Functional and Physical Assessment

Exercise Tolerance: Measured using the 6-Minute Walk Test (6MWT).

Physical Fitness and Strength: Assessed via Handgrip Dynamometry, the Barthel Scale for daily living activities, and the Tinetti Scale for balance and gait.

Body Composition: Detailed analysis using Bioelectrical Impedance Analysis (BIA) to track changes in muscle mass and fat tissue.

Diaphragm Function: Evaluation of diaphragm muscle thickness and mobility using Ultrasound (USG) to monitor respiratory improvement.

Postural Stability: Assessment of pressure distribution using a tensiometric mat (posturography).

B. Psychological and Neurocognitive Assessment

Mental Status: Evaluated using validated scales, including the WHO-5 Well-Being Index and the HADS Scale for anxiety and depression.

Cognitive Function: Screening for potential post-surgery cognitive impairment (memory, concentration) using the MoCA and MMSE scales.

C. Sleep Disorders and Biological/Hormonal Factors

Obstructive Sleep Apnea (OSA): Objective assessment of the frequency and severity of OSA using a portable sleep monitor.

Oral Health & OSA Risk: Detailed dental and craniofacial examinations to assess OSA risk factors related to the oral cavity status.

Hormonal and Biochemical Markers: Analysis of sex hormones (Testosterone, Estradiol) and their correlation with overall condition and rehabilitation response.

Myokines and Metabolic Signaling: Measurement of myokines (Irisin, Myostatin) and related proteins to understand mechanisms of exercise adaptation.

Standard Laboratory Tests: Including standard markers like lipid profile, glucose, HbA1c, CRP, homocysteine, and Vitamin D3.

Significance and Expected Outcomes The project aims to establish a patient profile that clearly identifies who benefits most from CR and who is at risk of poor outcomes. This identification of predictive factors will enable the early introduction of personalized interventions, such as targeted physical therapy, psychological support, or specialized diagnostics for sleep disorders. The ultimate goal is to optimize CR programs, maximizing gains in physical capacity, quality of life, and the long-term cardiac prognosis for patients.

ELIGIBILITY:
Inclusion Criteria:

* Male patients aged 50-80 years
* Hospitalization in the Cardiac Rehabilitation Ward
* Undergone coronary artery bypass graft (CABG) surgery within the last 30 days
* Written, informed consent to participate in the study

Exclusion Criteria:

* Type II diabetes treated with insulin
* Neuro-surgical operation in the last 6 months
* Aneurysms of the cerebral arteries and aorta
* Recurrent ischemic stroke (Cerebral Vascular Accident)
* Presence of a pacemaker
* Current treatment with testosterone

Ages: 50 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Male patients aged 50-80 years who have undergone coronary artery bypass graft (CABG) surgery and are currently hospitalized for cardiac rehabilitation. The study population includes individuals from a single clinical center in Poland.
Sampling Method: Non-Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2026-01-03 (Estimated); Primary Completion 2029-06-20 (Estimated); Study Completion 2029-07-01 (Estimated)

PRIMARY OUTCOMES:
Change in Physical Capacity (6MWT) | Baseline (start of hospitalization/T0) and Post-Rehab (end of cardiac rehabilitation/T1, approximately 3-4 weeks later)
  Distance walked in 6 minutes measured in meters using the 6-Minute Walk Test (6MWT). The test reflects objective functional improvement in physical capacity.

SECONDARY OUTCOMES:
Change in Psychological Status (HADS) | Baseline, Post-Rehab (approx. 3-4 weeks later), and Follow-up (3-6 months after discharge
  Assessment using the Hospital Anxiety and Depression Scale (HADS). The scale consists of 14 items (7 for anxiety and 7 for depression). Each item is scored from 0 to 3. Total score for each subscale ranges from 0 to 21. Higher scores indicate greater severity of anxiety or depression.
Diaphragm Thickness | Baseline and Post-Rehab (approx. 3-4 weeks later).
  Assessment of diaphragm muscle thickness measured in millimeters (mm) using Ultrasound (USG) at the end of expiration.
Change in Diaphragm Mobility | Baseline and Post-Rehab (approx. 3-4 weeks later).
  Assessment of diaphragm excursion measured in centimeters (cm) during maximum inspiration and expiration using Ultrasound (USG).
Change in Montreal Cognitive Assessment (MoCA) Score | Baseline, Post-Rehab (approx. 3-4 weeks later), and Follow-up (3-6 months after discharge).
  Cognitive screening using the MoCA scale. Total score ranges from 0 to 30. Higher scores indicate better cognitive function with a score of 26 or above generally considered normal.
Change in Mini-Mental State Examination (MMSE) Score | Baseline, Post-Rehab (approx. 3-4 weeks later), and Follow-up (3-6 months after discharge).
  Cognitive screening using the MMSE scale. Total score ranges from 0 to 30. Higher scores indicate better cognitive function where a score of 24-30 is typically considered normal.

OTHER OUTCOMES:
Change in Apnea-Hypopnea Index (AHI) | Baseline and Post-Rehab (approx. 3-4 weeks later).
  Frequency and severity of Obstructive Sleep Apnea (OSA) events assessed using a portable sleep monitor. The outcome is the number of apneas and hypopneas per hour of sleep (AHI index)
Change in Sex Hormones Concentration | Baseline (fasting) and Post-Rehab (fasting, approx. 3-4 weeks later)
  Serum concentration of Total Testosterone (measured in ng/dL) and Estradiol (measured in pg/mL).
Change in Myokines and Metabolic Markers Concentration | Baseline (fasting) and Post-Rehab (fasting, approx. 3-4 weeks later).
  Serum concentration of Irisin and Myostatin (measured in ng/mL) and other related markers (e.g., PGC-1α, FNDC5, mTOR)